CLINICAL TRIAL: NCT01085487
Title: MiCo - Mirena or Conventional Medical Treatment for Menorrhagia (MA0901)
Brief Title: MiCo - Mirena or Conventional Medical Treatment for Menorrhagia
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Global Medical Affairs Therapeutic Area Head, Bayer Healthcare
Other Study IDs: 14536; MA0901 (Other: company internal); MA0701-14697 (Other: company internal)
Record Dates: First submitted 2010-03-09; First posted 2010-03-12 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Idiopathic Menorrhagia
Keywords: Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1
  Interventions: Drug: Levonorgestrel (Mirena, BAY86-5028)
- Group 2
  Interventions: Drug: Hormonal treatment
- Group 3
  Interventions: Drug: Antifibrinolytic treatment

INTERVENTIONS:
Drug: Levonorgestrel (Mirena, BAY86-5028) — Women using Mirena for treatment of menorrhagia
  Groups: Group 1
Drug: Hormonal treatment — Hormonal treatment (including combined oral contraceptives or oral or injectable progestogens)
  Groups: Group 2
Drug: Antifibrinolytic treatment — Antifibrinolytic treatment (such as tranexamic acid)
  Groups: Group 3

SUMMARY:
The aim of this prospective, non-interventional post-marketing surveillance study is to obtain data on safety and efficacy of Mirena in treatment of heavy menstrual bleeding (Menorrhagia) under daily-life treatment conditions.For each patient, an initial visit and one to three follow-up visits after about 3, 6 and 12 months will be documented by the treating physician on the case report form. Observations include the patient's demographic parameters (date of birth, height, weight, race and smoking habits), previous contraceptives and menorrhagia treatment, gynaecological history, baseline menstruation, result of insertion, concomitant medications and diseases as well as menorrhagia symptoms. Overall treatment success will be evaluated at the end of treatment including number of weeks until improvement and reduction of menstrual bleeding with respect to duration and severity, and patient's satisfaction.

DETAILED DESCRIPTION:
The "MiCo - Mirena or conventional medical treatment for menorrhagia" study consist of two parts, MiCo Asia-Pacific and MiCo MA0901 (Rest of World).

Data from both parts will be analysed in separate pools as well as in a global pool. The trial alias are IMPACT Nos. 14697 (NCT00864136), 14536.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-45 (inclusive) not intending to become pregnant during the next year
* Women complaining of heavy menstrual bleeding over several consecutive cycles
* Women without structural or histological abnormality of the uterus, or with fibroids less than 3 cm in diameter which are causing no distortion of the uterine cavity (eligible for pharmaceutical treatment according to the NICE guideline 2007)
* Informed consent (where required by laws or regulations)

Exclusion Criteria:

* The contraindications and warnings of the respective Summary of Product Characteristics (Mirena®, combined oral contraceptives, oral/injectable progestogens, non-steroidal anti-inflammatory drug, or anti-fibrinolytic agent) must be followed.
* Women taking hormone replacement therapy
* Women with symptoms such as intermenstrual or post-coital bleeding, unless an endometrial biopsy has been performed and pathology excluded
* Women with fibroids that are palpable abdominally or who have intra-cavity fibroids and/or whose uterine length as measured at ultrasound or hysteroscopy is greater than 12 cm (NICE guideline 2007)
* Women on anticoagulative therapy or other treatment (including e.g. Copper IUD use) known to cause menorrhagia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 1211 (Actual)
Dates: Start 2009-04; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cumulative continuation rate at 12 months stratified by history of previous treatment(s) for menorrhagia | 12 months

SECONDARY OUTCOMES:
Bleeding pattern | 12 months
Patient satisfaction at end of documentation | 12 months
Impact of the therapy in terms of patient-reported health outcomes assessed using a validated questionnaire (Shaw RW et. al., British Journal of Obstetrics and Gynaecology, Vol 105(11), 1998.) | 12 months
Safety profile (adverse events) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Many Locations, Albania
- Many Locations, Bosnia and Herzegovina
- Many Locations, Colombia
- Many Locations, Croatia
- Many Locations, Czechia
- Many Locations, Jordan
- Many Locations, Lebanon
- Many Locations, Moldova
- Many Locations, North Macedonia
- Many Locations, Romania
- Many Locations, South Africa
- Many Locations, Syria
- Many Locations, Ukraine
- Many Locations, Venezuela